CLINICAL TRIAL: NCT02700282
Title: Impact of Backpack Position on Lung Function and Oxygen Consumption in School-aged Children With Cystic Fibrosis
Brief Title: Backpack Carrying in Children With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A01467-42
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Backpack carrying; Respiratory function; Children
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystic Fibrosis children (Experimental): Children with Cystic Fibrosis will experience lung function measurement while backpack carrying.
  Aerobic Capacities will also be assessed during treadmill gait.
  Interventions: Behavioral: Backpack Carrying
- Healthy Children (Active Comparator): Healthy Children will experience lung function measurement while backpack carrying.
  Aerobic Capacities will also be assessed during treadmill gait.
  Interventions: Behavioral: Backpack Carrying

INTERVENTIONS:
Behavioral: Backpack Carrying — A 12,5% of body weight backpack will be used for each measurement. Lung function will be assessed while carrying a double strap backpack, a mono shoulder backpack and without a backpack.

SUMMARY:
Cystic Fibrosis is a hereditary, chronic respiratory illness. Cystic Fibrosis leads to a progressive decline in lung function.

School-aged children with cystic fibrosis experience backpack carrying everyday. Backpack carrying induce a restrictive effect responsible for lower lung function. Respiratory muscle strength is also impaired.

No studies assessed aerobic capacities during children's gait while carrying a backpack.

The investigators hypothesized that backpack carrying will induce an acute decline in lung function in children with cystic fibrosis compared to healthy children. Investigators also hypothesized that aerobic capacities will be impaired.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis
* School-aged children (10 to 18)

Exclusion Criteria:

* Backpack carrying contraindication
* Acute exacerbation
* Impossible gait
* Other respiratory disease (asthma ...)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Lung Function (Forced Vital Capacity) | Immediate assessment while standing

SECONDARY OUTCOMES:
Lung function (Forced Expiratory Volume in 1 second) | Immediate assessment while standing
Respiratory Muscle Strength (MIP) | Immediate assessment while standing
  Maximal inspiratory pressure
Respiratory Muscle Strength (MEP) | Immediate assessment while standing
  Maximal expiratory pressure
Oxygen uptake (VO2) | During 12min treadmill gait
Ratio Ventilation/VO2 (Ventilation equivalent for oxygen) | During 12min treadmill gait
  Number of liters of air must be ventilated to consume 1 Liter of O2
Ratio Ventilation/VCO2 (Ventilation equivalent for carbon dioxide) | During 12min treadmill gait
  Number of liters of air must be ventilated to reject 1 Liter of CO2
Dyspnea (Borg Scale) | During 12min treadmill gait

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Le Roux, MD, Study Director — Le Havre Hospital
Locations (1):
- Le Havre Hospital, Le Havre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vieira AC, Ribeiro F. Impact of backpack type on respiratory muscle strength and lung function in children. Ergonomics. 2015;58(6):1005-11. doi: 10.1080/00140139.2014.997803. Epub 2015 Jan 13. PMID 25584722
- [Background] Dockrell S, Simms C, Blake C. Schoolbag carriage and schoolbag-related musculoskeletal discomfort among primary school children. Appl Ergon. 2015 Nov;51:281-90. doi: 10.1016/j.apergo.2015.05.009. Epub 2015 Jun 11. PMID 26154227
- [Background] Thobani A, Alvarez JA, Blair S, Jackson K, Gottlieb ER, Walker S, Tangpricha V. Higher mobility scores in patients with cystic fibrosis are associated with better lung function. Pulm Med. 2015;2015:423219. doi: 10.1155/2015/423219. Epub 2015 Feb 18. PMID 25789173
- [Background] Ramsey KA, Ranganathan S. Interpretation of lung function in infants and young children with cystic fibrosis. Respirology. 2014 Aug;19(6):792-9. doi: 10.1111/resp.12329. Epub 2014 Jun 19. PMID 24948040
- [Background] Pastre J, Prevotat A, Tardif C, Langlois C, Duhamel A, Wallaert B. Determinants of exercise capacity in cystic fibrosis patients with mild-to-moderate lung disease. BMC Pulm Med. 2014 Apr 30;14:74. doi: 10.1186/1471-2466-14-74. PMID 24884656